CLINICAL TRIAL: NCT00725127
Title: Chronotherapy with Low-dose Aspirin for Primary Prevention of Cardiovascular Events in Subjects with Impaired Fasting Glucose or Diabetes (CARING Study).
Brief Title: Chronotherapy with Low-dose Aspirin for Primary Prevention
Acronym: CARING
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Ramon C. Hermida, Professor, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CARING-2008/1; 2008-002669-30
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes
Keywords: Aspirin; Chronotherapy; Primary prevention; Impaired fasting glucose; Type 2 diabetes; Total mortality; Myocardial infarction; Stroke; Angina pectoris; Chronic kidney disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Myocardial Infarction; Stroke; Angina Pectoris; Renal Insufficiency, Chronic | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 100 mg/day ASA upon awakening.
  Interventions: Drug: aspirin
- 2 (Active Comparator): 100 mg/day ASA at bedtime
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: aspirin — 100 mg/day upon awakening for five years
  Other Names: Aspirin on awakening
  Arms: 1
Drug: aspirin — 100 mg/day at bedtime for five years
  Other Names: Aspirin at bedtime
  Arms: 2

SUMMARY:
Brief summary:

Aspirin (ASA) has been shown to provide marked benefits in primary and secondary prevention of cardiovascular events. Substantial evidence suggests that low-dose ASA therapy should also be used as a primary prevention strategy in men and women with diabetes who are at high cardiovascular risk. On the other hand, there is current evidence on the potential benefits of low-dose ASA therapy in subjects with impaired fasting glucose, including those with metabolic syndrome. Most important, previous laboratory animal and clinical trial research convincingly demonstrates administration time-dependent (with reference to circadian rhythms) effects of ASA. Thus, the effects of ASA upon lipoperoxides, b-adrenergic receptors, and blood pressure (BP) in clinically healthy subjects depend on the circadian timing of ASA administration. The administration-time-dependent influence of ASA on BP was previously demonstrated in a randomized trial on healthy women and other independent double-blind, randomized, placebo-controlled clinical trials conducted, first, on clinically healthy subjects, a second one on normotensive and hypertensive subjects, a third one on pregnant women at high risk for preeclampsia and a fourth one in previously untreated patients with mild hypertension. The findings of these BP studies are consistent; BP-lowering effect of low-dose ASA is achieved when administered at bedtime but not upon awakening.

In keeping with the chronopharmacological effects of ASA and the previous findings suggesting that ASA at low dose may exert a potential beneficial effect on BP, endothelium function and cardiovascular function, this prospective, randomized, parallel-arm study will investigate the potential influence of ASA on the primary prevention of cardiovascular, cerebrovascular and renal events in subjects with either impaired fasting glucose (≥ 100 mg/dl) or previous diagnosis of type 2 diabetes mellitus, who will receive low-dose ASA (100 mg/day) at different circadian times (upon awakening or at bedtime) in relation to their rest-activity cycle.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 50 years of age.
* Impaired fasting glucose (≥ 100 and < 126 mg/dl) in the last available blood test prior (≤ 3 months) to randomization, or diagnosis of type 2 diabetes prior to randomization.
* All subjects must have at randomization a conventional clinic systolic/diastolic BP < 160/100 mmHg.
* Informed consent to participate in the study prior to any study procedures.

Exclusion Criteria:

* Known or suspected contraindications, including history of allergy to ASA.
* Uncontrolled essential hypertension of Grade 2-3, i.e., systolic BP ≥ 160 mmHg and/or diastolic BP ≥ 100 mmHg before randomization.
* Evidence of a secondary form of hypertension, to include coarctation of the aorta, hyperaldosteronism, renal artery stenosis, or pheochromocytoma.
* Known Keith-Wagener grade III or IV hypertensive retinopathy.
* History of hypertensive encephalopathy, cerebrovascular event, transient ischemic cerebral attack, or myocardial infarction prior to randomization.
* Type 1 diabetes mellitus.
* History of heart failure.
* Second or third degree heart block without a pacemaker.
* Concomitant unstable angina pectoris.
* Concomitant potentially life threatening arrhythmia or symptomatic arrhythmia.
* Clinically significant valvular heart disease.
* Evidence of hepatic disease as determined by one of the following: ALT or AST values > 2 x UNL known before randomization, a history of hepatic encephalopathy, history of esophageal varices, or history of portocaval shunt.
* Diagnosis of chronic kidney disease prior to randomization.
* History of malignancy including leukemia and lymphoma (but not basal cell skin cancer), or any other severe, life-threatening disease within the past five years.
* Any previous history of a systemic autoimmune disease.
* History of drug or alcohol abuse within the last two years.
* Use of any disallowed concomitant medication.
* Inability to communicate and comply with all study requirements.
* Persons directly involved in the execution of this protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2008-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effects of awakening vs. bedtime 100 mg/day ASA administration in subjects with impaired fasting glucose or type 2 diabetes on primary prevention of cardiovascular, cerebrovascular and renal fatal, and non-fatal events. | Five years

SECONDARY OUTCOMES:
To evaluate the effects of awakening vs. bedtime 100 mg/day ASA administration on primary prevention of cardiovascular fatal and non-fatal events (including cardiovascular death, myocardial infarction, angina pectoris, and coronary revascularization). | Five years
To evaluate the effects of awakening vs. bedtime 100 mg/day ASA administration on primary prevention of cerebrovascular fatal and non-fatal events (including hemorrhagic stroke, ischemic stroke, and transient ischemic attack). | Five years
To evaluate the effects of awakening vs. bedtime 100 mg/day ASA administration on primary prevention of chronic kidney disease and/or congestive heart failure, and/or peripheral artery disease. | Five years
To demonstrate that 100 mg/day ASA at bedtime offers a similar safety profile than 100 mg/day ASA upon awakening | Five years
To demonstrate that compliance with 100 mg/day ASA at bedtime is similar to that with 100 mg/day ASA upon awakening. | Five years
To evaluate, for all previous objectives, potential gender differences in the benefits of low-dose ASA for primary prevention. | Five years
To evaluate, for all previous objectives, potential differences in the benefits of low-dose ASA for primary prevention between patients with and without diabetes. | Five years
To evaluate, for all previous objectives, potential differences in the benefits of low-dose ASA for primary prevention between subjects with and without metabolic syndrome. | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Ramon C Hermida, PhD, Study Director — University of Vigo
Locations (19):
- Spain (19):
  - CS Friol, Friol, Lugo
  - CS Fingoi, Lugo, Lugo
  - Complexo Hospitalario Universitario de Ourense, Ourense, Orense
  - CS A Estrada, A Estrada, Pontevedra
  - CS Baiona, Baiona, Pontevedra
  - CS Bueu, Bueu, Pontevedra
  - CS A Guarda, La Guardia, Pontevedra
  - CS Valmiñor, Nigrán, Pontevedra
  - CS Panxón, Nigrán, Pontevedra
  - CS Lerez, Pontevedra, Pontevedra
  - CS Tomiño, Tomiño, Pontevedra
  - Bioengineering & Chronobilogy Labs., University of Vigo, Vigo, Pontevedra
  - CS Calle Cuba, Vigo, Pontevedra
  - CS A Doblada, Vigo, Pontevedra
  - CS Coia, Vigo, Pontevedra
  - CS Sardoma, Vigo, Pontevedra
  - CS Teis, Vigo, Pontevedra
  - CS Vilaboa, Vilaboa, Pontevedra
  - CS San Roque, Vilagarcía de Arousa, Pontevedra

IPD SHARING:
Plan to Share IPD: Undecided